CLINICAL TRIAL: NCT07382856
Title: Effect of Low-intensity Aerobic Regular Activity on Heart Rate Variability in Type 1 Diabetes
Acronym: ELARA-T1D
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Banja Luka (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PAT1D2025
Record Dates: First submitted 2026-01-07; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 diabetes; Heart rate variability; Low-intensity physical activity
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The exercise group will consist of patients with type 1 diabetes who will perform low-intensity physical activity in the postprandial period five days per week over a one-year observation period.
  Interventions: Behavioral: low-intensity physical activity; Other: Intensive insulin therapy
- Control group (Active Comparator): Type 1 diabetes patients characterized by a sedentary lifestyle, defined as engaging in low-intensity physical activity less than five days per week.
  Interventions: Other: Intensive insulin therapy

INTERVENTIONS:
Behavioral: low-intensity physical activity — The exercise intervention consists of low-intensity physical activity (brisk walking) lasting 30-60 minutes, performed five times weekly. Participants will maintain a workload corresponding to Training Zone 2 over the course of the one-year follow-up.
  Arms: Experimental group
Other: Intensive insulin therapy — The patients with diabetes type 1 in Control group will be physical active (low-intensity physical activity) less than five days per week (not exceeding 30 minutes per activity).

SUMMARY:
A monocentric prospective randomized trial included 35 patients with Type 1 diabetes. Participants were randomized into two groups: Group A with the patients who engaged in low-intensity physical activity five days per week over a one-year observation period and Group B with the patients who engaged in physical activity less than five days per week. The study included three clinical visits: at baseline, at six months, and at one year. Assessments included cyclo-ergometry and body composition analysis during the baseline visit and at six-month visit, while 24-hour Holter monitoring was conducted at baseline and at the final visit. Biochemical parameters and microvascular complication risk assessments were performed at every visit.

DETAILED DESCRIPTION:
The ELARA-T1D study aims to investigate the impact of regular, long-standing low-intensity aerobic physical activity on heart rate variability (HRV) and cardiovascular autonomic neuropathy (CAN) in patients with Type 1 Diabetes Mellitus (T1DM). While physical activity is a cornerstone of diabetes management, fear of hypoglycemia and lack of specific guidelines often prevent patients from engaging in exercise. The mechanisms by which physical activity improves cardiovascular outcomes are not yet fully understood. This study focuses on reducing cardiovascular risk in T1DM through an unstructured low-intensity physical activity five days per week for 30-60 min per exercise, in training zone 2.

This is a randomized, parallel-assignment longitudinal study. Following a screening phase (0-4 months) to verify inclusion/exclusion criteria and baseline laboratory status, eligible participants had been randomized into two groups:

Experimental Group (Group A): Introduction of low-intensity aerobic activity five days per week for 30-60 minutes. The intensity is individually determined via spiroergometry to achieve training zone 2.

Control Group (Group B): Maintenance of previous sedentary or low-activity lifestyle (not exceeding 30 minutes, less than five days per week).

The physical activity protocol is monitored using heart rate tracking (Garmin watches) to ensure patients stay within the prescribed intensity zones.

Assessment of glycemic control using the ambulatory glucose profile (APG) was conducted using a Guardian 4 continuous glucose monitoring (CGM) system (Medtronic, Northridge, CA, USA).

The study evaluates the progression of Cardiovascular Autonomic Neuropathy (CAN) using the 24-hour Holter ECG monitoring to assess HRV

The assessment schedule is as follows:

Baseline (Month 0): Laboratory testing (CBC, UACR, HbA1c, BUN, eGFR, AST, ALT, CK, lipid profile), evaluation of microvascular complications, Cardiac ultrasound, HRV assessment ( 24h Holter), spiroergometry, evaluation of glycemic control using the ambulatory glucose profile (APG).

Follow-up (Months 6): Repeat laboratory testing, spiroergometry and APG to track changes in cardiovascular fitness and metabolic control.

Final visit (Months 12): Repeat laboratory testing, evaluation of microvascular complications, HRV assessment and APG to track changes in cardiac autonomic function and metabolic control.

In addition, all subjects underwent CT coronary angiography. Long-term follow-up: Continuous monitoring every 6 months up to 60 months to evaluate the long-term sustainability of the intervention's effects on cardiovascular health and chronic vascular complications Objectives The primary goal is to determine if consistent, low-intensity exercise can delay the onset of CAN or to prevent progression of incipient CAN and improve cardiovascular fitness.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Type 1Diabetes at least six months prior to study enrollment
* Male or female patients over 18 years
* Willingness to perform physical activity 5 days/week.
* Absence of heavy, chronic microvascular complications.
* Absence of established Cardiovascular neuropathy.
* Absence of established ASCVD.

Exclusion Criteria:

* Type 2 Diabetes
* Active engagement in professional sports
* Limb amputation
* Blindness
* Active malignancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2024-02-22 (Actual); Primary Completion 2026-02-22 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in Heart Rate Variability (HRV) parameters. | Twelve months from the baseline.
  Assessment of HRV as a marker for Cardiovascular Autonomic Neuropathy (CAN). The measurement tool is a 24-hour Holter ECG monitor. Specific parameters include the Standard Deviation of NN intervals (SDNN) and Root Mean Square of Successive Differences (RMSSD).
  Unit of Measure: Milliseconds (ms).

SECONDARY OUTCOMES:
Change in Peak Oxygen Consumption (VO2 peak) | Six months from the baseline.
  Evaluation of cardiovascular fitness through maximal exercise testing on a cycle ergometer (spiroergometry).
  Unit of Measure: milliliters per kilogram per minute (ml/kg/min).
Change in Time in Range (TIR). | Six and twelve months from the baseline.
  Assessment of glycemic control using the Guardian 4 Continuous Glucose Monitoring (CGM) system. TIR is defined as the percentage of time spent within the glucose range of 3.9-10.0 mmol/L. Unit of Measure: Percentage (%) of time.
Change in Urine Albumin-to-Creatinine Ratio (UACR). | Six months from the baseline.
  Assessment of renal microvascular function via laboratory urinalysis. Unit of Measure: milligrams per gram (mg/g).

CONTACTS AND LOCATIONS:
Locations (1):
- University Clinical Centre of the Republic of Srpska, Banja Luka, Bosnia and Herzegovina

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in our article (text, tables, figures, appendices) will be shared with researchers to achieve the aims of their approved proposals.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available beginning six month following publication of the final study results and will be available for up to three years.
Access Criteria: Data request should be submitted to the Principal Investigator. Data requestors will need to sign a data access agreement and provide a scientifically sound research proposal.

REFERENCES:
- [Background] Alarcon-Gomez J, Chulvi-Medrano I, Martin-Rivera F, Calatayud J. Effect of High-Intensity Interval Training on Quality of Life, Sleep Quality, Exercise Motivation and Enjoyment in Sedentary People with Type 1 Diabetes Mellitus. Int J Environ Res Public Health. 2021 Nov 30;18(23):12612. doi: 10.3390/ijerph182312612. PMID 34886337
- [Background] Italy. Corte Costituzionale. Judgment, 25 May 1987. Annu Rev Popul Law. 1987;14:38. PMID 12346712
- [Background] Wilson LC, Peebles KC, Hoye NA, Manning P, Sheat C, Williams MJA, Wilkins GT, Wilson GA, Baldi JC. Resting heart rate variability and exercise capacity in Type 1 diabetes. Physiol Rep. 2017 Apr;5(8):e13248. doi: 10.14814/phy2.13248. PMID 28420762
- [Background] Moser O, Zaharieva D, Adolfsson P, Battelino T, Bracken RM, Buckingham BA, Danne T, Davis EA, Dovc K, Forlenza GP, Gillard P, Hofer SE, Hovorka R, Jacobs PJ, Mader JK, Mathieu C, Norgaard K, Oliver NS, O'Neal DN, Pemberton J, Rabasa-Lhoret R, Sherr JL, Sourij H, Tauschmann M, Yardley JE, Riddell MC. The Use of Automated Insulin Delivery around Physical Activity and Exercise in Type 1 Diabetes: A Position Statement of the European Association for the Study of Diabetes (EASD) and the International Society for Pediatric and Adolescent Diabetes (ISPAD). Horm Res Paediatr. 2024 Dec 10:1-28. doi: 10.1159/000542287. Online ahead of print. PMID 39657609
- [Background] Riddell MC, Li Z, Gal RL, Calhoun P, Jacobs PG, Clements MA, Martin CK, Doyle Iii FJ, Patton SR, Castle JR, Gillingham MB, Beck RW, Rickels MR; T1DEXI Study Group. Examining the Acute Glycemic Effects of Different Types of Structured Exercise Sessions in Type 1 Diabetes in a Real-World Setting: The Type 1 Diabetes and Exercise Initiative (T1DEXI). Diabetes Care. 2023 Apr 1;46(4):704-713. doi: 10.2337/dc22-1721. PMID 36795053
- [Background] Riddell MC, Peters AL. Exercise in adults with type 1 diabetes mellitus. Nat Rev Endocrinol. 2023 Feb;19(2):98-111. doi: 10.1038/s41574-022-00756-6. Epub 2022 Oct 31. PMID 36316391
- [Background] Moser O, Zaharieva DP, Adolfsson P, Battelino T, Bracken RM, Buckingham BA, Danne T, Davis EA, Dovc K, Forlenza GP, Gillard P, Hofer SE, Hovorka R, Jacobs PG, Mader JK, Mathieu C, Norgaard K, Oliver NS, O'Neal DN, Pemberton J, Rabasa-Lhoret R, Sherr JL, Sourij H, Tauschmann M, Yardley JE, Riddell MC. The use of automated insulin delivery around physical activity and exercise in type 1 diabetes: a position statement of the European Association for the Study of Diabetes (EASD) and the International Society for Pediatric and Adolescent Diabetes (ISPAD). Diabetologia. 2025 Feb;68(2):255-280. doi: 10.1007/s00125-024-06308-z. PMID 39653802
- [Background] Colberg SR, Sigal RJ, Yardley JE, Riddell MC, Dunstan DW, Dempsey PC, Horton ES, Castorino K, Tate DF. Physical Activity/Exercise and Diabetes: A Position Statement of the American Diabetes Association. Diabetes Care. 2016 Nov;39(11):2065-2079. doi: 10.2337/dc16-1728. No abstract available. PMID 27926890
- [Background] Maran A, Pavan P, Bonsembiante B, Brugin E, Ermolao A, Avogaro A, Zaccaria M. Continuous glucose monitoring reveals delayed nocturnal hypoglycemia after intermittent high-intensity exercise in nontrained patients with type 1 diabetes. Diabetes Technol Ther. 2010 Oct;12(10):763-8. doi: 10.1089/dia.2010.0038. PMID 20807120
- [Background] Yardley JE, Sigal RJ, Kenny GP, Riddell MC, Lovblom LE, Perkins BA. Point accuracy of interstitial continuous glucose monitoring during exercise in type 1 diabetes. Diabetes Technol Ther. 2013 Jan;15(1):46-9. doi: 10.1089/dia.2012.0182. Epub 2012 Nov 8. PMID 23137050
- [Background] Tikkanen-Dolenc H, Waden J, Forsblom C, Harjutsalo V, Thorn LM, Saraheimo M, Elonen N, Rosengard-Barlund M, Gordin D, Tikkanen HO, Groop PH; FinnDiane Study Group. Frequent and intensive physical activity reduces risk of cardiovascular events in type 1 diabetes. Diabetologia. 2017 Mar;60(3):574-580. doi: 10.1007/s00125-016-4189-8. Epub 2016 Dec 24. PMID 28013340
- [Background] Zebrowska A, Hall B, Kochanska-Dziurowicz A, Janikowska G. The effect of high intensity physical exercise and hypoxia on glycemia, angiogenic biomarkers and cardiorespiratory function in patients with type 1 diabetes. Adv Clin Exp Med. 2018 Feb;27(2):207-216. doi: 10.17219/acem/66354. PMID 29521064
- [Background] Rahbar S, Naimi SS, Reza Soltani A, Rahimi A, Akbarzadeh Baghban A, Khorami N. Are Twenty-Four Sessions of Aerobic Exercise Sufficient for Improving Cardiac Parameters in Diabetes Mellitus? A Randomized Controlled Trial. J Tehran Heart Cent. 2018 Apr;13(2):43-51. PMID 30483312
- [Background] de Moraes R, Van Bavel D, Gomes MB, Tibirica E. Effects of non-supervised low intensity aerobic excise training on the microvascular endothelial function of patients with type 1 diabetes: a non-pharmacological interventional study. BMC Cardiovasc Disord. 2016 Jan 27;16:23. doi: 10.1186/s12872-016-0191-9. PMID 26817606
- [Background] Valletta JJ, Chipperfield AJ, Clough GF, Byrne CD. Daily energy expenditure, cardiorespiratory fitness and glycaemic control in people with type 1 diabetes. PLoS One. 2014 May 14;9(5):e97534. doi: 10.1371/journal.pone.0097534. eCollection 2014. PMID 24826899
- [Background] Serhiyenko VA, Serhiyenko AA. Cardiac autonomic neuropathy: Risk factors, diagnosis and treatment. World J Diabetes. 2018 Jan 15;9(1):1-24. doi: 10.4239/wjd.v9.i1.1. PMID 29359025
- [Background] Rohling M, Strom A, Bonhof GJ, Roden M, Ziegler D. Cardiorespiratory Fitness and Cardiac Autonomic Function in Diabetes. Curr Diab Rep. 2017 Oct 23;17(12):125. doi: 10.1007/s11892-017-0959-z. PMID 29063207
- [Background] Nystoriak MA, Bhatnagar A. Cardiovascular Effects and Benefits of Exercise. Front Cardiovasc Med. 2018 Sep 28;5:135. doi: 10.3389/fcvm.2018.00135. eCollection 2018. PMID 30324108
- [Background] Bohn B, Herbst A, Pfeifer M, Krakow D, Zimny S, Kopp F, Melmer A, Steinacker JM, Holl RW; DPV Initiative. Impact of Physical Activity on Glycemic Control and Prevalence of Cardiovascular Risk Factors in Adults With Type 1 Diabetes: A Cross-sectional Multicenter Study of 18,028 Patients. Diabetes Care. 2015 Aug;38(8):1536-43. doi: 10.2337/dc15-0030. Epub 2015 May 26. PMID 26015557
- [Background] Adu-Sarkodie NY. Clinical Management of Diabetes Mellitus in the Older Adult Patient. Curr Diabetes Rev. 2017;13(3):225-238. doi: 10.2174/1573399812666161206151706. PMID 27924723
- [Background] Pedersen BK, Saltin B. Exercise as medicine - evidence for prescribing exercise as therapy in 26 different chronic diseases. Scand J Med Sci Sports. 2015 Dec;25 Suppl 3:1-72. doi: 10.1111/sms.12581. PMID 26606383
- [Background] Pedersen BK. Which type of exercise keeps you young? Curr Opin Clin Nutr Metab Care. 2019 Mar;22(2):167-173. doi: 10.1097/MCO.0000000000000546. PMID 30640736